CLINICAL TRIAL: NCT00126308
Title: A Multi-Centre, Open-Label, Randomised Study to Assess the Efficacy, Durability and Safety of Immediate Versus Deferred Injections of Poly-L-Lactic Acid for HIV Facial Lipoatrophy (FLASH)
Brief Title: Facial Lipoatrophy Trial: Immediate Versus Deferred Injections of Poly-L-Lactic Acid for HIV Facial Lipoatrophy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no change in primary endpoint at week 48
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other); Abbott (Industry); Bristol-Myers Squibb (Industry); Gilead Sciences (Industry); GlaxoSmithKline (Industry); Merck Sharp & Dohme LLC (Industry); Hoffmann-La Roche (Industry); AIDS Council of New South Wales (Other)
Responsible Party: The National Centre in HIV Epidemiology and Clinical Research, The National Centre in HIV Epidemiology and Clinical Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V1-0 4-05; ACTR012605000132640
Record Dates: First submitted 2005-08-01; First posted 2005-08-03 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-03

CONDITIONS: HIV-Associated Lipodystrophy; HIV Infections
Keywords: HIV; Lipodystrophy; Intervention; Poly-L-lactic acid; HIV facial lipoatrophy; Treatment Experienced
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; HIV Infections; Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate (Experimental): poly-L-lactic acid injections
  Interventions: Device: poly-L-lactic acid
- Delayed (Active Comparator): poly-L-lactic acid injections
  Interventions: Device: poly-L-lactic acid

INTERVENTIONS:
Device: poly-L-lactic acid — immediate injections poly-L-lactic acid (4 bilateral treatments - 8 vials)
  Other Names: Sculptra
  Arms: Immediate
Device: poly-L-lactic acid — delayed (24 weeks) poly-L-lactic acid injections (4 bilateral treatment - 8 vials)
  Other Names: Sculptra
  Arms: Delayed

SUMMARY:
This is a multi-centre, open-label, 96 week study to evaluate the safety, tolerability and extent and duration of improvement in HIV-1 infected subjects with antiretroviral induced facial lipoatrophy, randomised in a 1:1 ratio to receive immediate or deferred deep subcutaneous injections of poly-L-lactic acid (PLA). Subjects will receive 4 treatments of PLA approximately every 2nd week, either at trial entry or following a delay period of 24 weeks.

DETAILED DESCRIPTION:
HIV lipodystrophy can be distressing and result in suboptimal antiretroviral (ART) adherence. Physical changes may stigmatise subjects while the negative psychological and social impact has become a major concern. To date, as there is no proven therapy for lipoatrophy, cosmetic interventions for facial lipoatrophy are being studied. Poly-L-lactic acid (PLA) has been shown to be both safe and effective when administered by injection to facial areas.

Study aims are:

1. to evaluate the extent and duration of improvement in HIV facial lipoatrophy of PLA injections;
2. to evaluate the impact of PLA injections on quality of life and ART adherence in subjects with HIV facial lipoatrophy;
3. to evaluate the safety and tolerability of polylactic acid.

100 HIV-infected ART-experienced subjects with facial lipoatrophy will be randomised in a 1:1 ratio at study entry to receive either immediate or deferred treatment (delayed 24 weeks) treatment with PLA. Randomisation will be stratified by age, severity of facial lipoatrophy, current ART (PI or non-PI containing and thymidine- or non-thymidine-containing) and surgeon.

The study has clinical end points monitoring CD4 cell counts, viral loads and adverse events. The study also has psychosocial end points monitoring quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more with laboratory evidence of HIV-1 infection
* Received combination antiretroviral therapy (minimum of 2 agents)
* Antiretroviral regimen should be stable for at least 12 weeks prior to entry with no changes planned during the first 48 weeks. For subjects not on antiretroviral therapy at entry there should be no intent to commence therapy in first 24 weeks.
* Moderate or severe facial lipoatrophy and lipodystrophy at one or more other sites
* Provide written, informed consent.

Exclusion Criteria:

* Active AIDS-defining illness including active HIV wasting
* Active herpes labialis or any acute or currently present chronic skin disease (infection/inflammation) on/near area to be treated
* Currently on anticoagulants or any coagulopathy that would preclude safe deep subcutaneous injections
* Women: pregnant, breastfeeding or have positive pregnancy test or not willing to use adequate contraception if of child-bearing potential
* Concomitant therapy with anabolic steroids (except testosterone replacement), corticosteroids at greater than replacement doses, growth hormone or any currently available or experimental agent to improve appetite or weight
* Testosterone replacement for less than 6 months or at greater than replacement doses
* Subjects who have discontinued any prohibited concomitant agent/s must cease this therapy at least 30 days prior to screening.
* Prior use of any facial dermal filling/tissue expansion agent/s
* Any condition which may interfere with ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint at 24 weeks will be change from baseline in facial soft tissue volume as measured by spiral computed tomography (CT). | 24 weeks

SECONDARY OUTCOMES:
Change from baseline at week 96 in facial soft tissue volume as measured by spiral CT scan | 96 weeks
Change from baseline at weeks 24 and 96 in physician and patient assessment of facial lipoatrophy severity | 24 and 96 weeks
Change from baseline at weeks 24 and 96 in peripheral fat as assessed by dual-energy X-ray absorptiometry (DEXA) | 24 and 96 weeks
Change from baseline at weeks 24 and 96 in quality of life | 24 and 96 weeks
Change from baseline at weeks 24 and 96 in antiretroviral therapy (ART) adherence and plasma HIV-RNA | 24 and 96 weeks
All serious, grade 3 or 4 clinical adverse events and any adverse event leading to change/s in ART or discontinuation of PLA | 24 and 96 weeks
All serious, grade 3 or 4 clinical adverse events (AEs) and any event leading to change/s in ART reported to week 96 | 96 weeks
All AEs attributable to study treatment reported to week 96 | week 96

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Carr, A/Prof, Principal Investigator — Immunology and Infectious Disease Unit, St. Vincent's Hospital, Sydney
Locations (18):
- Australia (18):
  - Dr Doong's Surgery, Burwood, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - 407 Doctors, Sydney, New South Wales
  - AIDS Research Initiative, Sydney, New South Wales
  - Albion Street Clinic, Sydney, New South Wales
  - Holdsworth House General Practice, Sydney, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Liverpool Health Service, Sydney, New South Wales
  - Waratah Clinic, St. George Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Queensland Health - AIDS Medical Unit, Brisbane, Queensland
  - Gladstone Road Medical Centre, Brisbane, Queensland
  - Gold Coast Sexual Health Clinic, Gold Coast, Queensland
  - Clinic 87, Nambour, Queensland
  - The Care and Prevention Programme - Adelaide University, Adelaide, South Australia
  - Royal Perth Hospital, Perth, Western Australia

REFERENCES:
- See also: NCHECR Website (Australia) — http://www.med.unsw.edu.au/nchecr/